CLINICAL TRIAL: NCT00873145
Title: Modular Prosthetic Reconstruction of Major Bone Defects of the Distal Humerus.
Brief Title: Management of Bone Defects Around the Elbow
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Philipp T. Funovics, Medical University of Vienna
Other Study IDs: funovics1
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2009-03

CONDITIONS: Tumor; Fracture; Cancer
Keywords: Survival; Function; Infection; Revision; Loosening
MeSH Terms: conditions — Neoplasms; Fractures, Bone; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with major bone defects around the elbow.
  Interventions: Procedure: HMRS

INTERVENTIONS:
Procedure: HMRS — Modular prosthetic replacement of the humerus and elbow.

SUMMARY:
Background:

Bone defects of the distal humerus require complex reconstructions, for which standard prostheses may be insufficient. The researchers therefore investigated the clinical and radiological outcome of elbow reconstructions by megaprostheses.

DETAILED DESCRIPTION:
Type of prosthesis:

STRYKER Humerus-HMRS

ELIGIBILITY:
Inclusion Criteria:

* HMRS of the elbow, distal humerus or total humerus

Exclusion Criteria:

* Unwillingness to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with major bone defects around the elbow and/or distal humerus due to cancer or failed arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Patient Survival | 20 Years

SECONDARY OUTCOMES:
Prosthetic Survival | 20 Years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna Department of Orthopaedics, Vienna, Austria